CLINICAL TRIAL: NCT06482164
Title: The THINK Study (Testing Hypoesthesia and the Incidence of Neurotrophic Keratopathy)
Brief Title: The THINK Study Incidence of Neurotrophic Keratopathy)
Acronym: THINK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20241252
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry Eye Disease (Other): Patients who have signs of dry eye
  Interventions: Diagnostic Test: Dry Eye Disease

INTERVENTIONS:
Diagnostic Test: Dry Eye Disease — Corneal sensitivity in patients who also have dry eye.

SUMMARY:
The study purpose is to evaluate corneal sensitivity in patients that have Stage 1 Neurotrphic Keratopathy (NK). Identifying patients with Stage 1 NK, may predict those who will in the future require rhNGF for optimal visual performance.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate corneal sensitivity in a cross-section of patients with signs of dry eye disease (DED), correlating findings against clinical parameters relating to the severity of disease and impact on quality of vision. Identifying those patients with Stage 1 Neurotrophic Keratopathy (NK), i.e. those with corneal staining and reduced sensitivity, may predict those who will in the future require rhNGF for optimal visual performance.

ELIGIBILITY:
Inclusion Criteria:

*Patients with the following: A diagnosis of dry eye disease Central or inferior corneal fluorescein staining defined by the Oxford Scale Reduced tear break up time (TBUT) ≤ 10 seconds.

* Able to comprehend and sign a statement of informed consent.
* Willing and able to complete all required postoperative visits.

Exclusion Criteria:

* Ocular surgery (e.g., intraocular, oculoplastic, corneal, or refractive surgical procedure) performed within the last 3 months or at any time in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Evidence of BAK or other chemical toxicity that, in the best judgment of the investigator, is causing reduced corneal sensitivity
* Concomitant use of daily contact lenses that, in the best judgment of the investigator, is causing reduced corneal sensitivity
* Clinically significant ocular trauma.
* Active ocular Herpes simplex or Herpes Zoster infection
* Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
* Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan, or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
* Active, systemic, or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the study findings.
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis.
* Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
* Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
* Participation in this trial in the same patient's fellow eye
* Patients who are under age 18, pregnant or breastfeeding, or who may become pregnant during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Patients with stage 1 neurotrophic keratopathy (NK) | Baseline Visit 0
  Patients with stage 1 neurotrophic keratopathy NK among dry eye patients

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Harvard Eye Associates
Locations (1):
- Harvard Eye Associates, Laguna Beach, California, United States